CLINICAL TRIAL: NCT04828499
Title: To Compare the Progressive Cracking Technique and Conventional Chop Technique on Corneal Endothelial Cells in Patients With Hard Nucleus Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WDD-hard-nucleus cataract
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Hard Nuclear Cataract; Corneal Endothelial Cell; Progressive Cracking Technique
MeSH Terms: interventions — Transcription Factor CHOP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Cracking Technique (Experimental): Patients with hard nucleus cataract were treated with Progressive Cracking Technique.
  Interventions: Procedure: Progressive Cracking Technique
- Conventional Chop Technique (Experimental): Patients with hard nucleus cataract were treated with Conventional Chop Technique.
  Interventions: Procedure: Conventional Chop Technique

INTERVENTIONS:
Procedure: Progressive Cracking Technique — Performing the cataract surgery with our phaco chop-progressive cracking technique.
  Arms: Progressive Cracking Technique
Procedure: Conventional Chop Technique — Performing the cataract surgery with Conventional Chop Technique.
  Other Names: stop and chop
  Arms: Conventional Chop Technique

SUMMARY:
Approximately 60 participants at Eye Hospital of Wenzhou Medical University during January,2017 to June 2021 will be enroll in our study. And dived them randomly into 2 groups:Progressive Cracking Technique (30 eyes) and Conventional Chop Technique (30 eyes) .

ELIGIBILITY:
Inclusion Criteria:

* Cataract with Grade IV~V nucleus sclerosis
* Cataract surgery is planned
* The operation was successful without any complications

Exclusion Criteria:

* Patients with other diseases that affect the corneal endothelium
* Has a history of anterior segment surgery
* Failure to cooperate with follow-up

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
corneal endothelial cell density | up to 1 months
  the number of corneal endothelial cells per unit area.
Coefficient of variation of endothelial cells | up to 1 months
  represents the variation coefficient of cell area
percentage of hexagonal cells of the cells marked | up to 1 months
  represents the percentage of hexagon cells,the ideal value is above 50%
central corneal thickness | up to 1 months
  thickness in micrometer

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided